CLINICAL TRIAL: NCT05267418
Title: Effects of Automated Oxygen Titration Alone or With High Flow Nasal Therapy on Dyspnea and Exercise Tolerance in Patients With Desaturating Chronic Lung Disease: a Randomized Clinical Trial
Brief Title: Effects of Automated Oxygen Titration Alone or With High Flow Nasal Therapy on Dyspnea and Exercise Tolerance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19 pandemia
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Francois Maltais, Principal Investigator, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21726
Record Dates: First submitted 2022-01-31; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Dyspnea; Lung Diseases; Pulmonary Hypertension; Chronic Obstructive Pulmonary Disease; Cystic Fibrosis; Interstitial Lung Disease
MeSH Terms: conditions — Dyspnea; Lung Diseases; Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant was not inform about what kind of oxygen support was provided during exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- automated nasal oxygen titration with FreeO2 alone (Active Comparator): The participant received automated nasal oxygen titration administered by a closed loop system (FreeO2) during the 3-min constant speed shuttle test (3-min CSST) and endurance shuttle walking test (ESWT). The objective of this system is maintain SpO2 a the pre-specified target level (94% in this study) with an automatic adjustment of oxygen flow second by second.
  Interventions: Device: Automated nasal O2 titration with FreeO2
- automated nasal oxygen titration with FreeO2 with high-flow nasal O2 therapy (Active Comparator): In addition to nasal oxygen titration administered by a closed loop system (FreeO2), the participant received high flow nasal therapy (Airvo2) set at 60 liters per minute with nasal canula during the 3-min CSST and endurance shuttle walking test.
  Interventions: Device: Automated nasal O2 titration with FreeO2
- Fixed-flow oxygen therapy (Active Comparator): The participant received oxygen by nasal canula at a fixed flow of 2 liters per minute during the 3-min constant speed shuttle test (3-min CSST) and endurance shuttle walking test (ESWT). In patients already on home oxygen, the O2 flow during exercise was set at 1 L/min above the usual flow used at home .
  Interventions: Device: Automated nasal O2 titration with FreeO2

INTERVENTIONS:
Device: Automated nasal O2 titration with FreeO2 — The participant received, in a randomized, cross-over study design: 1) automated nasal oxygen titration administered by a closed loop system (FreeO2) alone, 2) or with high flow nasal therapy (Airvo2) set at 60 liters per minute with nasal canula, or 3) oxygen by nasal canula at a fixed flow of 2 liters per minute during the 3-min constant speed shuttle test (3-min CSST) and endurance shuttle walking test (ESWT)
  Other Names: High O2 nasal flow with Airvo2; Fixed O2 flow

SUMMARY:
The main purpose of this study is to evaluate the effects of automated oxygen administration (FreeO2 system) alone or with high-flow oxygen on dyspnea and exercise tolerance in people with desaturating chronic lung disease compared to fixed oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

One of them

* Moderate to severe COPD (forced expiratory volume in 1 second (FEV1) < 80% predicted and FEV1/forced vital capacity (FVC) ratio < 0.7)
* Chronic interstitial lung disease such as usual interstitial pneumonitis (UIP), non-specific interstitial pneumonitis (NSIP) or hypersensitivity pneumonitis on high-resolution computed tomography
* Pulmonary arterial hypertension type 1 or 4, excluding involvement secondary to collagenosis as well as secondary to congenital heart disease, as diagnosed with mean pulmonary artery pressure > 25 mm Hg at right heart catheterization
* Cystic fibrosis, as diagnosed by a positive sweat test (>60 mmol/L) or having 2 genetic mutations known to cause cystic fibrosis.

AND having a 6-minute walking test with significant desaturation defined as a decrease in O2 saturation greater or equal to 5% with O2 saturation at the end of the walking test < 88%

Exclusion Criteria:

* Exacerbation of the primary lung disease in the past 8 weeks
* Exercise limiting diseases other than the primary lung disease.
* Not reaching the target dyspnea score during the walking tests.
* Stage 1 pulmonary sarcoidosis
* History of syncope on exertion
* SpO2 with effort less than 90% despite the use of 6 L of O2 per minute
* Cardiac condition deemed unstable or severe (e.g. severe aortic stenosis)
* Disabling or severe rheumatological or neurological condition
* Participation in a pulmonary rehabilitation program within the last year
* Patients with multi-resistant bacteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Dyspnea score | At the end of the 3 minute-constant speed shuttle test (CSST) (3 minutes), immediately after the intervention (either fixed-O2, automated nasal O2 adjustment alone, or automated nasal O2 adjustment + high nasal flow)
  Dyspnea score on the modified Borg scale (0 to 10, with higher score indicating worse dyspnea)

SECONDARY OUTCOMES:
Endurance time duration of the Endurance Shuttle Walking Test (EWST) | Duration in (mm:ss) of Endurance Shuttle Walking Test (ESWT), immediately after the intervention (either fixed-O2, automated nasal O2 adjustment alone, or automated nasal O2 adjustment + high nasal flow)
  Total duration of Endurance Shuttle Walking Test
Mean pulsed O2 saturation (SpO2) during Endurance Shuttle Walking Test (EWST) | From the beginning to the end of the Endurance Shuttle Walking Test (ESWT) which will be done on 3 testing days, with either fixed O2, automatic O2 adjustment alone, or automatic O2 adjustment + high nasal flow
  Mean % pulsed O2 saturation (SpO2) during the Endurance Shuttle Walking Test (ESWT)

OTHER OUTCOMES:
Mean pulsed O2 saturation (SpO2) during 3min-CSST | From the beginning to the end of the 3 minute-constant speed shuttle test which will be done on 3 testing days with either fixed O2, automatic O2 adjustment alone, or automatic O2 adjustment + high nasal flow)
  The mean % pulsed O2 saturation (SpO2) during the test duration time
Capillary blood gases | Difference the baseline capillary PCO2 from the resting values (before Endurance Shuttle Walking Test - ESWT) to the end of exercise values (after the Endurance Shuttle Walking Test - ESWT) immediately after the intervention
  Carbon dioxide partial pressure (PCO2), lactate

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Background] Maltais F, Aumann JL, Kirsten AM, Nadreau E, Macesic H, Jin X, Hamilton A, O'Donnell DE. Dual bronchodilation with tiotropium/olodaterol further reduces activity-related breathlessness versus tiotropium alone in COPD. Eur Respir J. 2019 Mar 28;53(3):1802049. doi: 10.1183/13993003.02049-2018. Print 2019 Mar. PMID 30655277
- [Background] Beaulieu J, Jensen D, O'Donnell DE, Brouillard C, Tracey L, Vincent S, Nadreau E, Bernard E, Bernard S, Maltais F. Relieving exertional dyspnea during the 3-min constant speed shuttle test in patients with COPD with indacaterol/glycopyrronium versus tiotropium: the RED trial. Ther Adv Respir Dis. 2020 Jan-Dec;14:1753466620939507. doi: 10.1177/1753466620939507. PMID 32663102
- [Background] Perrault H, Baril J, Henophy S, Rycroft A, Bourbeau J, Maltais F. Paced-walk and step tests to assess exertional dyspnea in COPD. COPD. 2009 Oct;6(5):330-9. doi: 10.1080/15412550903156317. PMID 19863362